CLINICAL TRIAL: NCT05279859
Title: A Phase 1b/2 Master Protocol of Agents Targeting the Mitogen-Activated Protein Kinase Pathway in Patients With Hematologic Malignancies
Brief Title: A Study of Anti-Cancer Therapies Targeting the MAPK Pathway in Patients With Hematologic Malignancies
Acronym: HERKULES-4
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-007-04
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; FLT3; mutation; relapsed; refractory; gilteritinib; Xospata; MAPK; SHP2; ERK
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Part 1): ERAS-007 plus gilteritinib (Experimental): ERAS-007 will be administered in combination with gilteritinib to study participants with R/R FLT3 mutated AML in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: Gilteritinib
- Dose Escalation (Part 2): ERAS-601 plus gilteritinib (Experimental): ERAS-601 will be administered in combination with gilteritinib to study participants with R/R FLT3 mutated AML in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-601; Drug: Gilteritinib
- Dose Expansion (Part 3): ERAS-007 plus gilteritinib (Experimental): ERAS-007 will be administered at the recommended dose (as determined from Part 1) in combination with gilteritinib to study participants with R/R FLT3 mutated AML.
  Interventions: Drug: ERAS-007; Drug: Gilteritinib
- Dose Expansion (Part 4): ERAS-601 plus gilteritinib (Experimental): ERAS-601 will be administered at the recommended dose (as determined from Part 2) in combination with gilteritinib to study participants with R/R FLT3 mutated AML.
  Interventions: Drug: ERAS-601; Drug: Gilteritinib

INTERVENTIONS:
Drug: ERAS-007 — Administered orally
  Arms: Dose Escalation (Part 1): ERAS-007 plus gilteritinib; Dose Expansion (Part 3): ERAS-007 plus gilteritinib
Drug: ERAS-601 — Administered orally
  Arms: Dose Escalation (Part 2): ERAS-601 plus gilteritinib; Dose Expansion (Part 4): ERAS-601 plus gilteritinib
Drug: Gilteritinib — Administered orally
  Other Names: Xospata

SUMMARY:
* To evaluate the safety and tolerability of escalating doses of ERAS-007 or ERAS-601 in combination with other cancer therapies in study participants with hematologic malignancies.
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-007 or ERAS-601 administered in combination with other cancer therapies.
* To evaluate the preliminary efficacy of ERAS-007 or ERAS-601 in combination with other cancer therapies in study participants with hematologic malignancies.
* To evaluate the PK profiles of ERAS-007 or ERAS-601 and other cancer therapies when administered in combination.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, multicenter master protocol evaluating safety, tolerability, and preliminary efficacy of ERAS-007 or ERAS-601 in combination with other cancer therapies in study participants with hematologic malignancies. The study will commence with dose escalation cohorts (ERAS-007 plus gilteritinib and ERAS-601 plus gilteritinib) in study participants with relapsed or refractory (R/R) Feline McDonough sarcoma (FMS)-like tyrosine kinase 3 (FLT3) mutated acute myeloid leukemia (AML). Dose expansion will follow and will evaluate ERAS-007 or ERAS-601 drug combinations administered at the RD identified from each respective dose escalation cohort in study participants with R/R FLT-3 mutated AML.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willing and able to give written informed consent.
* Diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) according to World Health Organization classification.
* Relapsed after or refractory to first-line AML therapy.
* Positive for FLT3 mutation in bone marrow or whole blood.
* Eastern Cooperative Oncology Group performance status ≤ 2 with no deterioration during screening period.
* Adequate hepatic and renal function.
* Recovery from non-hematologic AEs associated with prior therapy to baseline CTCAE v5 Grade 0 or 1, except for AEs not considered a safety risk (eg, alopecia or vitiligo).
* Able to take oral medication with no medical conditions that prevent swallowing and absorbing oral medications.
* Willing to comply with all protocol-required visits, assessments, and procedures.

Exclusion Criteria:

* Diagnosis of AML secondary to prior chemotherapy or other neoplasms (except for MDS).
* Diagnosis of acute promyelocytic leukemia or BCR-ABL-positive leukemia (chronic myeologenous leukemia in blast crisis).
* Clinically active central nervous system leukemia.
* Second or later hematologic relapse or prior salvage therapy for refractory disease.
* For participants being considered for ERAS-007+gilteritinib treatment: prior therapy with ERK inhibitor.
* For participants being considered for ERAS-601+gilteritinib treatment: prior therapy with SHP2 inhibitor.
* Anticancer therapy ≤14 days prior to first dose (except hydroxyurea given for controlling blast count), or ≤5 half-lives prior to first dose, whichever is shorter.
* Palliative radiation ≤7 days prior to first dose.
* Major surgery within 28 days of enrollment.
* Contraindication to gilteritinib use as per local label.
* Known hypersensitivity to any of the components of ERAS-007 or ERAS-601.
* Clinically active infection, requiring systemic therapy.
* Impaired cardiovascular function or clinically significant cardiovascular disease.
* History of thromboembolic or cerebrovascular events ≤6 months prior to first dose.
* History of other malignancy ≤3 years prior to first dose.
* History of retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vein occlusion (RVO), or risk factors to RPED or RVO.
* History of or clinically active interstitial lung disease (ILD), drug induced ILD, or radiation pneumonitis that required steroid treatment.
* Any evidence of severe or uncontrolled systemic disease or evidence of any other significant clinical disorder or laboratory finding that renders the participant inappropriate to participate in the study.
* Pregnant or breastfeeding women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Maximum Tolerated Dose (MTD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Recommended Dose (RD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma concentration of ERAS-007 or ERAS-601 and other cancer therapies
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma concentration of ERAS-007 or ERAS-601 and other cancer therapies
Area under the curve | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve of ERAS-007 or ERAS-601 and other cancer therapies
Half-life | Study Day 1 up to Day 29
  Half-life of ERAS-007 or ERAS-601 and other cancer therapies
Antileukemic activity | Assessed up to 24 months from time of first dose
  Percentage of Participants With Complete Remission and Complete Remission With Partial Hematological Recovery (CR/CRh); CR rate
Duration of antileukemic activity | Assessed up to 24 months from time of first dose
  Duration of CR/CRh (DOCR/DOCRh)
Duration of antileukemic activity | Assessed up to 24 months from time of first dose
  Duration of CR (DOCR)

CONTACTS AND LOCATIONS:
Overall Officials: Les Brail, Ph.D., Study Director — Medical Monitor
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Texas Oncology, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No